CLINICAL TRIAL: NCT05462964
Title: The Effect of the Use of Pacifier and Pacifier With Dextrose on Reducing Pain During Orogastric Tube Insertion in Newborns: A Randomized Controlled Trial
Brief Title: Reducing Pain During Orogastric Tube Insertion in Newborns: Use of Pacifiers and Pacifiers Sweetened With 25% Dextrose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Aysenur Akkaya Gul, Lecturer, Uludag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UludagUniversity-AKKAYAGUL
Record Dates: First submitted 2022-07-04; First posted 2022-07-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Pain
Keywords: Neonatal; Orogastric tube; Pacifiers; %25 Dextrose; NIPS
MeSH Terms: conditions — Pain | interventions — Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): Newborns in this group were started to camera recording 2 minutes before the procedure and routine OGT placement was performed. It was checked whether the orogastric tube was in the right place. After the evaluation period was completed and the baby was comfortable, the recording was stopped.After OGT insertion, a light touch was provided if necessary to ensure routine comfort of the baby for ethical reasons.
- İntervention Group 1 (Experimental): Only a pacifier was given to the newborn.
  Interventions: Behavioral: Pacifiers Group (İntervention Group 1)
- İntervention Group 2 (Experimental): The newborn was given a pacifier sweetened with 25% dextrose.
  Interventions: Behavioral: Pacifier group sweetened with 25% dextrose (İntervention Group 2)

INTERVENTIONS:
Behavioral: Pacifiers Group (İntervention Group 1) — Camera recording was started 2 minutes before OGT placement and only a pacifier was given to the newborn. After the pacifier in the OGT intervention group was placed in the mouth of the given baby in the form of leaking from the mouth, it was inserted by advancing the baby's swallowing reflex from the esophagus to the stomach. It was checked whether the orogastric tube was in the right place. After the evaluation period was completed and the baby was comfortable, the recording was stopped.
  Arms: İntervention Group 1
Behavioral: Pacifier group sweetened with 25% dextrose (İntervention Group 2) — Camera recording was started 2 minutes before OGT insertion and the newborn was given a pacifier sweetened with 25% dextrose. After the dextrose-sweetened pacifier in the OGT intervention group was placed in the mouth of the baby in the form of a leak from the mouth, it was inserted by advancing the baby's esophagus and then to the stomach with the swallowing reflex of the baby. It was checked whether the orogastric tube was in the right place. After the evaluation period was completed and the baby was comfortable, the registration was stopped.
  Arms: İntervention Group 2

SUMMARY:
Orogastric tube(OGT) placement, which is used for monitoring, diagnostic and therapeutic purposes, causes pain and stress in premature and term newborns. Non-pharmacological pain intervention with pacifiers and sweetener solutions (sucrose, dextrose, etc.) in newborns is a viable nursing approach to reduce pain. In the limited number of studies in the literature, it was seen that pacifiers and sucrose were used in nasogastric tube(NGT) applications and they were especially focused on premature babies. In our study, due to the fact that it was conducted in term newborns and, unlike the limited number of studies, OGT was placed in the stomach in the form of a pacifier and a 25% dextrose pacifier leaking from the rim. Our study was conducted as a randomized controlled experimental study to examine the effect of using pacifiers and dextrose pacifiers on pain reduction during orogastric tube placement, and also to evaluate the effects on behavioral response and physiological parameters (heart rate, oxygen saturation) in newborns.In addition, it was thought that the fact that the study was carried out by passing a pacifier and a pacifier sweetened with 25% dextrose, would facilitate progress and reduce trauma by stimulating the swallowing reflex in newborns via a pacifier as in adults.The population of the study consisted of term newborns at 38-42 weeks of gestation who were hospitalized in the Neonatal Intensive Care Unit of a hospital in Turkey between April-December 2019. The sample group randomly consisted of 60 newborns (Control group: 20, Intervention group with only pacifiers:20, with dextrose flavored pacifiers:20). 20 babies in the intervention group were given only pacifiers and 20 babies were given a pacifiers flavored with dextrose 2 minutes before the OGT insertion. The procedure was performed by leaking the tube from the edge of the pacifiers. Routine OGT insertion was performed in the control group. The data collection process was recorded with a camera. The Neonatal Infant Pain Scale (NIPS), the highest heart rate and lowest oxygen saturation from physiological pain responses, and crying time from behavioral parameters were evaluated by the researcher by watching the camera recording. Variance analysis, Shapiro Wilk, Kruskal Wallis, Chi-square, Bonferro, and Wilcoxon tests were used in the statistical analysis of the study. The SPSS v22 package program was used for statistical analysis and the significance level was taken at α=0.05.

DETAILED DESCRIPTION:
Painful and invasive procedures for follow-up, diagnostic and therapeutic purposes are an inevitable part of care in the neonatal intensive care unit. Effective pain management is at the core of nursing care and is based on a comprehensive assessment of the infant and its pain. Nurses and the interdisciplinary healthcare team have a responsibility to prevent or minimize pain during these procedures. Studies to reduce pain during OGT insertion were generally performed in premature newborns, but there are few studies performed in term newborns. It has been observed that there are not enough studies on OGT that focus on NGT placement in the studies. In the studies examined, the use of dextrose and pacifier alone, which are non-pharmacological methods in reducing pain, were generally discussed, and no studies involving the combined use were found. It is thought that our study will be useful in terms of the fact that feeding tube placement, which is known to be a painful and stressful procedure, will be performed in term newborns, presenting new evidence to nurses for reducing pain and stress, and supporting the existing study results.

This study is a randomized controlled experimental study to examine the effect of using pacifiers and dextrose pacifiers on pain reduction during orogastric tube placement in newborns, as well as to evaluate behavioral responses and physiological changes in newborns. In addition, it was thought that the fact that the study was carried out by passing a pacifier and a pacifier sweetened with 25% dextrose, would facilitate progress and reduce trauma by stimulating the swallowing reflex in newborns via a pacifier as in adults. Ethical approval was obtained from the Bursa Uludağ University Faculty of Medicine Clinical Research Ethics Committee before starting the study. In order to start the research after the approval of the ethics committee, T.C. Permissions were obtained from the Istanbul Provincial Health Directorate and the Istanbul Tuzla State Hospital management. In addition, written consent was obtained from the families of the newborns in the control and intervention groups, with an informed consent form. The research was carried out in Turkey/Istanbul Tuzla State Hospital neonatal intensive care unit between April-December 2019. The population consisted of term newborns who were hospitalized in the neonatal intensive care unit of Istanbul Tuzla State Hospital, whose OGT placement procedure was deemed clinically appropriate, and legal permission was obtained from their families. Of these newborns, a total of 60 newborns, 20+20 in the intervention group and 20 in the control group, were included in the sample group. The first intervention group consisted of 20 newborns given a pacifier alone, the second intervention group consisted of 20 newborns given a pacifier sweetened with 25% dextrose, and 20 newborns in the control group. Randomization was provided by the researcher for babies who met the inclusion criteria of the study during weekday neonatal intensive care unit working hours. For this; During working hours, the first newborn to be fitted with OGT was in the control group, the second newborn was given a pacifier only, and the third newborn was in the pacifier intervention group sweetened with 25% dextrose. When there was not enough OGT indication (less than 3) on the same day, the application continued in the same order in the next clinical shift. It was applied in the same way for each group before the procedure. Information about the baby and the mother in the baby and mother introduction form, which was prepared by using the literature, was filled in before the procedure. The newborns were placed under a radiant warmer in an open bed 5 minutes before the procedure. In newborns who could not be placed under a radiant heater, the application was performed in an incubator. After the preparation of the necessary materials before the application, the OGT measurement to be placed was made and the marking process was carried out. A saturation probe was placed in the baby to monitor heart rate and oxygen saturation. The newborn was prepared for the procedure by adjusting the camera monitor focused on the baby's face in the field of view. 2 minutes before OGT insertion, 20 babies in the intervention groups were given pacifiers alone, and 20 babies were given pacifiers sweetened with 25% dextrose. The procedure was carried out by leaking the tube from the pacifiers. In the control group, routine OGT placement was performed without giving anything. The data collection process was recorded with a camera. After the evaluation period was completed and the baby was comfortable, the recording was stopped. However, the recording continued without any time constraint to monitor the crying time of the baby who continued to cry during the insertion. The dependent variables of the study were the score from the NIPS pain scale, oxygen saturation, heart rate, and crying time.

ELIGIBILITY:
Inclusion Criteria:

* Babies are term newborns with 38-42 weeks of gestation,
* Having a newborn for whom only OGT insertion will be attempted,
* Having a newborn who did not receive any painful stimuli until 30 minutes before the intervention,
* The parent's volunteering for the newborn to participate in the study formed the inclusion criteria.

Exclusion Criteria:

* Newborns with any congenital anomalies of the face or oral cavity,
* Newborns with 3rd and 4th degree intraventricular hemorrhage,
* Newborns receiving muscle relaxants, analgesics, and sedation formed the exclusion criteria of the study.

Ages: 38 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2018-12-25 (Actual); Primary Completion 2020-02-18 (Actual); Study Completion 2020-02-18 (Actual)

PRIMARY OUTCOMES:
Neonatal Infant Pain Scale (NIPS) | Pre-procedure
  The Neonatal Infant Pain Scale (NIPS) scale was used for pain assessment.The primary outcome was the pain score assessed with NIPS scale, a validated and widely used tool to measure procedural pain in infants. NIPS is a measurement tool that includes five behavioral groupings (facial expression, crying, movements of arms and legs, state of alertness) and one physiological parameter (respiration pattern). Of the indicators, only crying is scored between 0 and 2, while the other indicators are scored as 0 or 1. Evaluation results in a possible total score between 0 and 7. A high score indicates an increase in the severity of pain.NIPS pain assessment: pre-procedure, during the procedure, 1st minute and 3rd minute after OGT placement.
Neonatal Infant Pain Scale (NIPS) | During the procedure
  The Neonatal Infant Pain Scale (NIPS) scale was used for pain assessment.The primary outcome was the pain score assessed with NIPS scale, a validated and widely used tool to measure procedural pain in infants. NIPS is a measurement tool that includes five behavioral groupings (facial expression, crying, movements of arms and legs, state of alertness) and one physiological parameter (respiration pattern). Of the indicators, only crying is scored between 0 and 2, while the other indicators are scored as 0 or 1. Evaluation results in a possible total score between 0 and 7. A high score indicates an increase in the severity of pain.NIPS pain assessment: pre-procedure, during the procedure, 1st minute and 3rd minute after OGT placement.
Neonatal Infant Pain Scale (NIPS) | 1st minute after OGT placement.
  The Neonatal Infant Pain Scale (NIPS) scale was used for pain assessment.The primary outcome was the pain score assessed with NIPS scale, a validated and widely used tool to measure procedural pain in infants. NIPS is a measurement tool that includes five behavioral groupings (facial expression, crying, movements of arms and legs, state of alertness) and one physiological parameter (respiration pattern). Of the indicators, only crying is scored between 0 and 2, while the other indicators are scored as 0 or 1. Evaluation results in a possible total score between 0 and 7. A high score indicates an increase in the severity of pain.NIPS pain assessment: pre-procedure, during the procedure, 1st minute and 3rd minute after OGT placement.
Neonatal Infant Pain Scale (NIPS) | 3rd minute after OGT placement.
  The Neonatal Infant Pain Scale (NIPS) scale was used for pain assessment.The primary outcome was the pain score assessed with NIPS scale, a validated and widely used tool to measure procedural pain in infants. NIPS is a measurement tool that includes five behavioral groupings (facial expression, crying, movements of arms and legs, state of alertness) and one physiological parameter (respiration pattern). Of the indicators, only crying is scored between 0 and 2, while the other indicators are scored as 0 or 1. Evaluation results in a possible total score between 0 and 7. A high score indicates an increase in the severity of pain.NIPS pain assessment: pre-procedure, during the procedure, 1st minute and 3rd minute after OGT placement.

SECONDARY OUTCOMES:
Highest Heart Rate | Within 15 seconds before OGT insertion
  Nellcor Bedside Console Type Pulse Oximeter Device was used to monitor heart rate. The recording was made by adjusting the camera focused on the baby's face to show the pulse oximeter device within the field of view. Highest heart rate was evaluated from camera recordings within 15 seconds before OGT insertion, during the procedure, and at 3 minutes after insertion.
Highest Heart Rate | During the procedure
  Nellcor Bedside Console Type Pulse Oximeter Device was used to monitor heart rate. The recording was made by adjusting the camera focused on the baby's face to show the pulse oximeter device within the field of view. Highest heart rate was evaluated from camera recordings within 15 seconds before OGT insertion, during the procedure, and at 3 minutes after insertion.
Highest Heart Rate | 3 minutes after insertion
  Nellcor Bedside Console Type Pulse Oximeter Device was used to monitor heart rate. The recording was made by adjusting the camera focused on the baby's face to show the pulse oximeter device within the field of view. Highest heart rate was evaluated from camera recordings within 15 seconds before OGT insertion, during the procedure, and at 3 minutes after insertion.
Lowest Oxygen Saturation | Within 15 seconds before OGT insertion
  Nellcor Bedside Console Type Pulse Oximeter Device was used to monitor heart rate. The recording was made by adjusting the camera focused on the baby's face to show the pulse oximeter device within the field of view. The lowest oxygen saturation was evaluated from camera recordings within 15 seconds before OGT insertion, during the procedure, and at 3 minutes after insertion.
Lowest Oxygen Saturation | During the procedure
  Nellcor Bedside Console Type Pulse Oximeter Device was used to monitor heart rate. The recording was made by adjusting the camera focused on the baby's face to show the pulse oximeter device within the field of view. The lowest oxygen saturation was evaluated from camera recordings within 15 seconds before OGT insertion, during the procedure, and at 3 minutes after insertion.
Lowest Oxygen Saturation | 3 minutes after insertion
  Nellcor Bedside Console Type Pulse Oximeter Device was used to monitor heart rate. The recording was made by adjusting the camera focused on the baby's face to show the pulse oximeter device within the field of view. The lowest oxygen saturation was evaluated from camera recordings within 15 seconds before OGT insertion, during the procedure, and at 3 minutes after insertion.
Crying Time | During the procedure
  Focusing on the baby's face, the camera also records sound. During the procedure, the recording continued without time constraint to monitor the crying time of the baby. The crying time during the procedure was evaluated by listening to the camera recording audibly.

CONTACTS AND LOCATIONS:
Locations (1):
- Uludag University, Bursa, Nilufer, Turkey (Türkiye)

REFERENCES:
- [Derived] Akkaya-Gul A, Ozyazicioglu N. Effect of pacifier and pacifier with dextrose in reducing pain during orogastric tube insertion in newborns: a randomized controlled trial. J Perinatol. 2024 May;44(5):717-723. doi: 10.1038/s41372-024-01948-w. Epub 2024 Mar 29. PMID 38553602